CLINICAL TRIAL: NCT02129751
Title: A Double-Blind, Placebo-Controlled, Multicenter Study of Efficacy and Safety of Bupropion Hydrobromide in Adolescents and Children With Major Depressive Disorder
Brief Title: Efficacy and Safety of Bupropion Hydrobromide in Adolescents and Children With Major Depressive Disorder
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-BUPA-401
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
Keywords: able to swallow medications without difficulty; bupropion hydrobromide
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- bupropion hydrobromide (Experimental): study drug
  Interventions: Drug: bupropion hydrobromide
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bupropion hydrobromide — study drug
  Other Names: Aplenzin
  Arms: bupropion hydrobromide
Drug: Placebo — placebo arm
  Arms: placebo

SUMMARY:
Double-Blind, Placebo-Controlled, Multicenter Study of Efficacy and Safety

DETAILED DESCRIPTION:
* The primary efficacy endpoint is the mean change from Baseline to EOT in total CDRS-R (raw) score.
* The secondary efficacy endpoints include:

  * Proportion of subjects characterized as responders at EOT (≥40% improvement from Baseline total CDRS-R raw score)
  * Proportion of subjects characterized as in remission at EOT (total CDRS-R raw score <29)
  * Mean change from Baseline to EOT in CGI-C.

Safety endpoints include:

* Incidence of AEs
* Change from Baseline to EOT in vital signs (blood pressure and radial pulse rate), blood and urine laboratory panel, and ECG
* Treatment discontinuation due to AEs
* Suicidality as assessed by the C-SSRS score
* Change from Baseline to EOT in sleep as assessed by the sleep subscale of the CDRS-R.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged ≥7 to <18 years (at Screening Visit 1).
* Provide assent (subject) and written informed consent (parent/legal representative) and Health Insurance Portability and Accountability Act (HIPAA) for study participation (at Screening Visit 1).
* Meet diagnostic criteria for MDD as defined in the DSM IV-TR5 at Screening Visits 1 and 1a (K-SADS-PL; see Appendix 17.2).
* Current depressive episode of at least 4 weeks' duration as noted in the subject's history (Screening Visit 1).
* Total CDRS-R raw score ≥45 at both the Screening and Baseline Visits (Visits 1 and 2) (see Appendix 17.3).
* CGI-S score of ≥4 at the Baseline Visit (Visit 2) (see Appendix 17.4).

Exclusion Criteria:

* are unable to swallow medications without difficulty
* have known hypersensitivity to bupropion hydrobromide
* are pregnant or planning to get pregnant or are lactating
* Women of childbearing age unable to use at least one method of effective contraception for the duration of the study
* Previous history of attempted suicide
* are unable to understand and communicate effectively with parent, Investigator, and study coordinator
* are at immediate risk of requiring hospitalization, in the Investigator's opinion
* have current seizure disorder or history of seizures or head trauma
* have history or presence of clinically significant medical conditions or clinically important laboratory abnormalities
* have ECG or physical examination abnormality at screening
* have body weight less than the 3rd percentile or greater than the 97th percentile for age.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline to EOT in total CDRS-R (raw) score | Baseline and 2 years
  Change from Baseline to EOT in total Children's Depression Rating Scale - Revised (CDRS-R). A higher score indicates a more profound state of depression. The interviewer rates 17 symptom areas; the symptom scores are summed to generate a total score. The total score ranges from 17 to 108.

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health